CLINICAL TRIAL: NCT07157774
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Effect of Muvalaplin on the Reduction of Major Adverse Cardiovascular Events in Adults With Elevated Lipoprotein(a) Who Have Had a Prior Atherosclerotic Cardiovascular Event or Are at Risk for a First Atherosclerotic Cardiovascular Event
Brief Title: Assessing the Impact of Muvalaplin on Major Cardiovascular Events in Adults With Elevated Lipoprotein(a)
Acronym: MOVE-Lp(a)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27269; 2025-521067-13-00 (EU CTIS Number); J2O-MC-EKBG (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Elevated Lp(a); Atherosclerotic Cardiovascular Disease (ASCVD)
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Muvalaplin (Experimental): Participants will receive muvalaplin orally.
  Interventions: Drug: Muvalaplin
- Placebo (Placebo Comparator): Participants will receive placebo orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Muvalaplin — Administered orally
  Other Names: LY3473329
  Arms: Muvalaplin
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of muvalaplin in reducing cardiovascular risk in participants with high lipoprotein(a) who have cardiovascular disease or are at risk of a heart attack or stroke.

ELIGIBILITY:
Inclusion Criteria:

* Have Lp(a) ≥175 nanomoles per liter (nmol/L)
* Meet one of the following criteria:

  * Have had a prior atherosclerotic cardiovascular disease (ASCVD) event (such as heart attack, stroke, or procedure to restore blood flow to the heart or other parts of the body) within 10 years prior to screening
  * Are at risk for a first ASCVD event, defined as one or more of the following:

    * Documented coronary artery disease (CAD), carotid stenosis, or peripheral artery disease (PAD) without a history of ASCVD event
    * A high coronary artery calcium (CAC) score
    * Reduced kidney function with diabetes
    * Combination(s) of high risk factors

Exclusion Criteria:

* Have experienced a major cardiovascular event or surgery, such as heart attack, stroke, or procedure to restore blood flow to the heart or other parts of the body, within 90 days prior to screening or occurring between screening and randomization
* Are planning or expected to undergo a procedure to restore blood flow in the arteries or a major heart surgery during the study
* Have uncontrolled high blood pressure
* Have New York Heart Association (NYHA) class III or IV heart failure
* Have undergone a procedure to remove cholesterol from the blood within 90 days of screening, or have a planned procedure during the study
* Have severe kidney impairment
* Have had cancer within 5 years prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10450 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2031-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Time to First Occurrence of Any Component of the Major Adverse Cardiac Event (MACE)-4 Composite Endpoint | Baseline up to End of Study (About 5.25 Years)
  Time to first event in a MACE-4 composite endpoint, comprised of cardiovascular death, nonfatal myocardial infarction, nonfatal ischemic stroke, and urgent coronary revascularization.

SECONDARY OUTCOMES:
Percent Change from Baseline in Lipoprotein(a) (Lp(a)) at Week 4 | Baseline, Week 4
Time to First Occurrence of Any Component of the MACE-3 Composite Endpoint | Baseline up to End of Study (About 5.25 Years)
Time to First Occurrence of Any Component of the Modified MACE-3 Composite Endpoint | Baseline up to End of Study (About 5.25 Years)
Time to First Occurrence of Any Component of the Coronary MACE-3 Composite Endpoint | Baseline up to End of Study (About 5.25 Years)
Time to First Occurrence of Any Component of MACE-3 + Major Adverse Limb Event (MALE) Composite Endpoint | Baseline up to End of Study (About 5.25 Years)
Time to Occurrence of All-Cause Mortality | Baseline up to End of Study (About 5.25 Years)
Time to First Occurrence of Each Individual Component of the MACE-4 Composite Endpoint | Baseline up to End of Study (About 5.25 Years)
Change from Baseline to Each Annual Visit for Health-Care Resource Utilization (HCRU) | Baseline up to End of Study (About 5.25 Years)
Pharmacokinetics (PK): Trough Concentration at Steady State (C-trough, ss) of Muvalaplin | Predose through Week 96

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (697):
- United States (80):
  - Prime Medical Group, LLC dba Gilbert Center for Family Medicine, LLC, Gilbert, Arizona
  - Axsendo Clinical Research - Peak Heart & Vascular - Phoenix, Phoenix, Arizona
  - Clinical Research Institute of Arizona (CRI) - Sun City West, Sun City West, Arizona
  - Southwest Kidney Institute - Surprise, Surprise, Arizona
  - Pima Heart, Tucson, Arizona
  - National Heart Institute, Beverly Hills, California
  - John Muir Medical Center - Concord Campus, Concord, California
  - Neighborhood Healthcare Institute of Health, Escondido, California
  - Ark Clinical Research - Fountain Valley, Fountain Valley, California
  - The Cardiovascular Center, Redding, California
  - UCLA South Bay Endocrinology, Torrance, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Legacy Clinical Trials, Colorado Springs, Colorado
  - OptumCare Clinical Trials, LLC, Golden, Colorado
  - FWD Clinical Research, Boca Raton, Florida
  - American Research Institute, Cutler Bay, Florida
  - Arrow Clinical Trials, Daytona Beach, Florida
  - Soffer Health Institute, Hollywood, Florida
  - K2 MEDICAL Research THE VILLAGES, Lady Lake, Florida
  - K2 Medical Research ORLANDO, Maitland, Florida
  - Dade Florida Clinical Research Center, Miami, Florida
  - Onhealth Research Center, Miami, Florida
  - Masters of Clinical Research, Augusta, Georgia
  - Elite Clinical Trials, Blackfoot, Idaho
  - CARE Institute - High Desert, Meridian, Idaho
  - Elite Clinical Trials, Rexburg, Idaho
  - Tulane University School of Medicine, New Orleans, Louisiana
  - MaineHealth Cardiology, Scarborough, Maine
  - Ascension Saint Agnes Heart Care, Baltimore, Maryland
  - Metropolitan Cardiovascular Consultants, Beltsville, Maryland
  - Johns Hopkins University, Columbia, Maryland
  - Centennial Medical Group, Columbia, Maryland
  - Anderson Medical Research, Ft. Washington, Maryland
  - Lucida Clinical Trials, New Bedford, Massachusetts
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - Boeson Research MSO, Missoula, Montana
  - Clinical Research of South Nevada, Las Vegas, Nevada
  - Vector Clinical Trials, Las Vegas, Nevada
  - Vector Clinical Trials, Sparks, Nevada
  - IMA Clinical Research, Albuquerque, New Mexico
  - Southwest Cardiovascular Center, Albuquerque, New Mexico
  - Capital Cardiology Associates, Albany, New York
  - NYC Research, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Rochester Clinical Research, LLC, Rochester, New York
  - Southgate Medical Group, West Seneca, New York
  - Kaiser Permanente Sunnyside Medical Center, Clackamas, Oregon
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - M3 Wake Research - Charleston, Charleston, South Carolina
  - Circle Clinical Research, Sioux Falls, South Dakota
  - WR-Clinsearch, LLC, Chattanooga, Tennessee
  - The Jackson Clinic, Jackson, Tennessee
  - PharmaTex Research, Amarillo, Texas
  - St. David's Heart & Vascular PLLC dba Austin Heart, Austin, Texas
  - Southwest Family Medicine Associates, Dallas, Texas
  - Renal Disease Research Institute, Dallas, Texas
  - IntraCare, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Texas Health Research & Education Institute - Fort Worth, Fort Worth, Texas
  - Cedar Health Research - Fort Worth, Fort Worth, Texas
  - GMG Clinical Research (DBA Radiance Clinical Research) - Lampasas, Lampasas, Texas
  - Revival Research Institute, LLC, McKinney, Texas
  - PRX Research, Mesquite, Texas
  - Sherman Clinical Research, Sherman, Texas
  - Ogden Clinic - Canyon View, Ogden, Utah
  - Advanced Research Institute, Ogden, Utah
  - Virginia Heart, Falls Church, Virginia
  - Mary Washington Hospital, Fredericksburg, Virginia
  - Carient Heart & Vascular - Manassas, Manassas, Virginia
  - Manassas Clinical Research Center, Manassas, Virginia
  - TPMG (Tidewater Physicians Multispecialty Group) Clinical Research, Newport News, Virginia
  - York Clinical Research, Norfolk, Virginia
  - Dominion Medical Associates, Inc., Richmond, Virginia
  - Carilion Clinic, Roanoke, Virginia
  - ERA Health Research - CardioNow - Lynnwood, Lynnwood, Washington
  - Eastside Research Associates, Redmond, Washington
  - Rainier Clinical Research Center, Renton, Washington
  - Universal Research Group, Tacoma, Washington
  - Central Washington Health Services Association d/b/a Confluence Health, Wenatchee, Washington
- Argentina (54):
  - CEC - Consultorios de Especialidades Cardiovasculares, Bahía Blanca
  - CONEXA Investigacion Clinica S.A., Buenos Aires
  - Buenos Aires Macula S.A, Buenos Aires
  - CIPREC, Buenos Aires
  - Kynet, Buenos Aires
  - Instituto Médico Especializado (IME), Buenos Aires
  - Consultorio Medico Dr Litvak Bruno, Buenos Aires
  - Cardiología Palermo, Buenos Aires
  - Consultorio Medico Investigador Principal Dr Besada, Buenos Aires
  - Glenny Corp. S.A., Buenos Aires
  - Stat Research S.A., Buenos Aires
  - Investigaciones Medicas Imoba Srl, Buenos Aires
  - Centro de Investigaciones Metabólicas (CINME), Buenos Aires
  - Mautalen Salud e Investigación, Buenos Aires
  - Consultorio de Investigación Clínica EMO SRL, Buenos Aires
  - CEMEDIC, Buenos Aires
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Buenos Aires
  - Fundación Respirar, Buenos Aires
  - Centro Médico Arsema, Buenos Aires
  - CEMEDIAB, C.a.b.a.
  - IDIM - Instituto de Investigaciones Metabólicas, Ciudad de Buenos Aires
  - Instituto de Cardiología "Juana F. Cabral", Corrientes
  - Instituto de Investigaciones Clínicas Córdoba, Córdoba
  - Centro Médico Colón, Córdoba
  - Centro Medico Privado San Vicente Diabetes, Córdoba
  - CIPADI - Centro Integral de Prevencion y Atencion en Diabetes, Godoy Cruz
  - Centro de Investigaciones Clínicas Baigorria, Granadero Baigorria
  - CMD-Centro Médico y Diagnóstico por Imágenes, Junín
  - CIMeL, Lanús
  - Polo de Salud Vistalba, Luján de Cuyo
  - Centro de Investigaciones Médicas Mar del Plata, Mar del Plata
  - Instituto de Investigaciones Clínicas Mar del Plata, Mar del Plata
  - Fundacion Scherbovsky, Mendoza
  - Instituto de Cardiología Wolff, Mendoza
  - Instituto De Investigaciones Clinicas Quilmes, Quilmes
  - DIM Clínica Privada, Ramos Mejía
  - Instituto Médico Río Cuarto, Río Cuarto
  - Centro Rosarino de Investigaciones Clinicas (CRICs), Rosario
  - Fundacion Estudios Clinicos, Rosario
  - INECO Neurociencias Oroño, Rosario
  - Instituto Especialidades de la Salud Rosario, Rosario
  - Instituto Médico Catamarca IMEC, Rosario
  - Instituto de Investigaciones Clinicas Rosario, Rosario
  - Laboratorio de Hemostasia y Trombosis, Rosario
  - Hospital Provincial del Centenario, Rosario
  - Santa Maria de la Salud Centro Medico, San Isidro
  - Corporación Médica San Martín, San Martín
  - Centro Modelo de Cardiología, San Miguel de Tucumán
  - Investigaciones Clínicas Tucumán, San Miguel de Tucumán
  - Centro de Diagnóstico y Rehabilitación (CEDIR), Santa Fe
  - Centro de Investigaciones Clinicas del Litoral, Santa Fe
  - Centro de Salud e Investigaciones Médicas, Santa Rosa
  - Centro de Investigaciones Medicas Temperley, Temperley
  - Instituto de Investigaciones Clinicas Zarate, Zárate
- Australia (15):
  - Nightingale Research, Adelaide
  - Box Hill Hospital, Box Hill
  - Royal Brisbane and Women's Hospital, Brisbane
  - Heart of Australia, Brisbane
  - Advara HeartCare - Burwood, Burwood
  - Victorian Heart Hospital, Clayton
  - Barwon Health, Geelong
  - Royal Hobart Hospital, Hobart
  - Ipswich Hospital, Ipswich
  - Sydney Cardiometabolic Centre, Liverpool
  - The AIM Centre / Hunter Diabetes Centre, Merewether
  - Advara HeartCare - Milton, Milton
  - Fusion Clinical Research, Norwood
  - Southern Adelaide Diabetes & Endocrine Services, Oaklands Park
  - Latrobe Regional Health, Traralgon
- Austria (18):
  - Krankenhaus St. Josef Braunau, Braunau am Inn
  - VIVIT, Feldkirch
  - Medizinische Universität Graz, Graz
  - Ordensklinikum Linz GmbH Elisabethinen, Linz
  - Konventhospital der Barmherzigen Brüder Linz, Linz
  - Cardio Metabolic Centre, Mattersburg
  - Landesklinikum Mistelbach, Mistelbach
  - Uniklinikum Salzburg, Salzburg
  - imed St. Pölten, Sankt Pölten
  - Universitätsklinikum St. Pölten, Sankt Pölten
  - Klinik Landstraße, Vienna
  - Zentrum für klinische Studien Dr Hanusch Gmbh, Vienna
  - Medizinische Universität Wien, Vienna
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna
  - Klinik Hietzing, Vienna
  - Herz Zentrum Währing - Innere Medizin und Kardiologie | Alle Kassen und Privat, Vienna
  - Imed19-privat, Vienna
  - Klinik Floridsdorf, Vienna
- Belgium (26):
  - AZORG Campus Aalst-Moorselbaan, Aalst
  - ANIMA Research, Alken
  - ZAS Middelheim, Antwerp
  - Imelda General Hospital, Bonheiden
  - Algemeen Ziekenhuis klina, Brasschaat
  - AZ Sint-Jan Brugge-Oostende AV, Bruges
  - Centre Hospitalier Universitaire Brugmann, Brussels
  - Cliniques universitaires Saint-Luc, Brussels
  - Antwerp University Hospital, Edegem
  - Ziekenhuis Oost-Limburg, Campus St.-Jan, Genk
  - Jan Yperman Ziekenhuis, Ieper
  - Kormont, Kluisbergen
  - AZ Groeninge Campus Kennedylaan, Kortrijk
  - UZ Leuven, Leuven
  - Clinical Chc Montlégia, Liège
  - InoKura, Liège
  - Gezondheidshuis De Gloed, Machelen
  - AZ Sint-Maarten, Mechelen
  - Meclinas, Mechelen
  - Pneumocare, Namur
  - AZ Oostende vzw, Ostend
  - Artsen Netwerk De Schelde, Oudenaarde
  - Artsenpraktijk OHIO, Oudenaarde
  - AZ Delta vzw, Roeselare
  - Private Practice - Dr. De Watertoren, Tielt
  - Private Practice - Dr. Tim Decraecke (Zwalm), Zwalm
- Brazil (38):
  - Centro de Pesquisa Clinica do Coracao, Aracaju
  - Hospital Universitário João de Barros Barreto, Belém
  - NUPEC - Cardio, Belo Horizonte
  - AngioKormann Blumenau, Blumenau
  - Hospital Sirio Libanes, Brasília
  - Hospital do Coração do Brasil, Brasília
  - Chronos Pesquisa Clínica, Brasília
  - Instituto de Pesquisa clinica de Campinas, Campinas
  - Centro de Pesquisa Sao Lucas, Campinas
  - Quanta Diagnóstico e Terapia, Curitiba
  - Instituto de Ensino e Pesquisa Clinica do Ceara, Fortaleza
  - Universidade Federal de Goias, Goiânia
  - C-MEP - Centro Multidisciplinar de Ensino e Pesquisa, Joinville
  - CPHOSP Manaus Medicina, Ensino e Pesquisa, Manaus
  - Instituto Do Coracao De Marilia, Marília
  - Instituto Atena de Pesquisa Clinica, Natal
  - Instituto Méderi de Pesquisa e Saúde, Passo Fundo
  - Hospital Maternidade E Pronto Socorro Santa Lucia, Poços de Caldas
  - Hospital de Clinicas de Porto Alegre, Porto Alegre
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre
  - Núcleo de Pesquisa Clínica do Rio Grande do Sul, Porto Alegre
  - Hospital Moinhos de Vento, Porto Alegre
  - Hospital Nossa Senhora da Conceição, Porto Alegre
  - Rede AME SAÚDE, Recife
  - Centro de Pesquisa Silvestre Santé, Rio Branco
  - IBPClin - Instituto Brasil de Pesquisa Clínica, Rio de Janeiro
  - Ruschel Medicina e Pesquisa Clínica, Rio de Janeiro
  - Inovace Pesquisa Clínica, Salvador
  - Praxis Pesquisa Medica, Santo André
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto
  - Centro Internacional de Pesquisa Clínica (CIPES), São José dos Campos
  - CPQuali Pesquisa Clínica, São Paulo
  - CPCLIN, São Paulo
  - Instituto Dante Pazzanese de Cardiology, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica, São Paulo
  - Incor - Instituto do Coracao, São Paulo
  - CEDOES, Vitória
  - Integral Pesquisa e Ensino, Votuporanga
- Canada (18):
  - Ecogene-21, Chicoutimi
  - Viacar Recherche Clinique, Greenfield Park
  - Winterberry Research Inc., Hamilton
  - Premier Clinical Trial Network, Hamilton
  - Diex Recherche Inc. Division Joliette, Joliette
  - G A Research Associates, Moncton
  - Institut de Cardiologie de Montreal, Montreal
  - North York Diagnostic and Cardiac Centre, North York
  - IUCPQ, Québec
  - Bluewater Clinical Research Group Inc., Sarnia
  - KMH Cardiology Centres - Stoney Creek, Stoney Creek
  - Unity Health Toronto, St. Michael's Hospital, Toronto
  - Riverside Cardiology and Diagnostic Imaging, Toronto
  - Diex Recherche Inc. Division Trois-Rivieres, Trois-Rivières
  - Victoria Heart Institute Foundation, Victoria
  - Discovery Clinical Services, Victoria
  - Fadia El Boreky Medicine, Waterloo
  - Clinical Research Solutions - Kitchener, Waterloo
- China (44):
  - Peking University First Hospital, Beijing
  - Xuanwu Hospital Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - Beijing Pinggu District Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - China-Japan Union Hospital, Changchun
  - Changde First People's Hospital, Changde
  - Xiangya Hospital Central South University, Changsha
  - The First People's Hospital of Changzhou, Changzhou
  - Sichuan Provincial People's Hospital, Chengdu
  - West China Hospital Sichuan University, Chengdu
  - 2nd Affiliated Hospital Chongqing Medical Universi, Chongqing
  - Daqing People's Hospital, Daqing
  - The First People's Hospital of Foshan, Foshan
  - Guangdong Provincial People's Hospital, Guangzhou
  - Zhujiang Hospital, Guangzhou
  - Zhejiang Hospital, Hangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - The First Hospital of Harbin Medical University, Harbin
  - The Second People's Hospital of Hefei, Hefei
  - Jinan Central Hospital, Jinan
  - Jining No.1 People's Hospital, Jining
  - Huaihe Hospital of Henan University, Kaifeng
  - Lishui Central Hospital, Lishui
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang Shi
  - Affiliated Hospital of Luzhou Medical College, Luzhou
  - Jiangxi Provincial People's Hospital, Nanchang
  - Nanchang People's Hospital, Nanchang
  - Zhongda Hospital Southeast University, Nanjing
  - Jiangsu Province Hospital, Nanjing
  - The first affiliated hospital of Ningbo university, Ningbo
  - Zhongshan Hospital,Fudan University, Shanghai
  - Shanghai Xuhui Central Hospital, Shanghai
  - The First Affiliated Hospital of Shantou University Medical College, Shantou
  - Siping Central People's Hospital, Siping
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - Chongqing Three Gorges Central Hospital, Wanzhou
  - The 2nd Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou
  - Renmin Hospital of Wuhan University, Wuhan
  - Shaanxi provincial people's hospital, Xi'an
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou
  - Xuzhou Central Hospital, Xuzhou
  - Zigong First People's Hospital, Zigong
- Czechia (17):
  - Kardiologie Stříbrný, Brno
  - MUDr. Karel Kamenik - Kardiologicka Ambulance, Brno
  - Kardiologická ambulance Brno, Brno
  - Kardio Chlumec, Chlumec nad Cidlinou
  - INTENDIA klinika s.r.o., Chrudim III
  - DR. HAUS - Kardiologicka Ambulance, Český Krumlov
  - DIKa Centrum, Havířov
  - CTC Hodonin s.r.o., Hodonín
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Cévní ambulance Nový Jičín, Nový Jičín
  - MUDr. Buchta s.r.o., Kardiologicka ambulance, Ostrava
  - Pratia Pardubice a.s., Pardubice
  - Diabet2 s.r.o., diabetologicka a interni ambulance, Prague
  - Clinoxus, Prague
  - Angiocentrum Komorany, Prague
  - Poliklinika Lípa Centrum, Prague
  - Cardio Research, s.r.o, Zlín
- Denmark (3):
  - Sanos Clinic - Nordjylland, Gandrup
  - Sanos Clinic, Herlev
  - Sanos Clinic - Syddanmark, Vejle
- France (16):
  - Centre Hospitalier Universitaire Dijon Bourgogne - Hôpital François Mitterrand, Dijon
  - Centre Hospitalier d'Annecy, Epagny Metz-Tessy
  - Chu Grenoble Alpes, La Tronche
  - Hopital Claude Huriez - CHU de Lille, Lille
  - Centre Hospitalier Saint Joseph - Saint Luc, Lyon
  - Hôpital Nord Guillaume-et-René-Laennec / CHU de Nantes, Nantes
  - Centre Hospitalier Universitaire de Nice - Hopital Pasteur, Nice
  - Pitie Salpetriere University Hospital, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Bichat - Claude-Bernard, Paris
  - Hôpital Saint Antoine, Paris
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Centre Hospitalier Universitaire de Saint Étienne - Hôpital Nord, Saint-Priest-en-Jarez
  - CHU Strasbourg-Hautepierre, Strasbourg
  - CHU Rangueil, Toulouse
  - Centre Hospitalier Régional Universitaire de Tours - Hôpital Bretonneau, Tours
- Germany (38):
  - Universitätsklinikum Aachen, Aachen
  - Zentrum für klinische Studien Bad Homburg, Bad Homburg
  - Klinische Forschung Berlin-Mitte, Berlin
  - Kardiologische Praxen im Spreebogen, Berlin
  - FutureMeds GmbH, Berlin
  - Charité Campus Virchow-Klinikum, Berlin
  - Klinische Forschung Dresden, Dresden
  - Zentrum für klinische Prüfungen in der Facharztzentrum Dresden-Neustadt Betriebsgesellschaft mbH, Dresden
  - Hausärztlich-Kardiologisches MVZ am Felsenkeller GmbH/Zentrum für klinische Studien, Dresden
  - Herzzentrum Dresden GmbH Universitätsklinik, Dresden
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden
  - Unterfrintroper Hausarztzentrum Klinische Forschung, Essen
  - Cardioangiologisches Centrum Bethanien, Frankfurt
  - ClinPhenomics CVC GmbH, Frankfurt
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Nephrologisches Zentrum Göttingen, Göttingen
  - Universitätsmedizin Greifswald, Greifswald
  - HRF II - Hamburger Rheuma Forschungszentrum II MVZ für Rheumatologie und Autoimmunmedizin Hamburg GmbH / -T, Hamburg
  - Klinische Forschung Hamburg, Hamburg
  - Cardiologicum Hamburg, Hamburg
  - Velocity Clinical Research, Hamburg, Hamburg
  - Klinische Forschung Hannover-Mitte, Hanover
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Klinische Forschung Karlsruhe, Karlsruhe
  - Universitätsklinikum Leipzig, Leipzig
  - Herzzentrum Leipzig GmbH, Leipzig
  - Universität zu Lübeck - Institut für Endokrinologie und Diabetes, Lübeck
  - Praxis Oedeme, Lüneburg
  - Otto-von-Guericke-Universität Magdeburg, Magdeburg
  - ze:ro ARZTPRAXEN, Mannheim
  - Deutsches Herzzentrum München, Munich
  - Institut für Diabetesforschung GmbH Münster, Münster
  - Dedicated Research Site FutureMeds, Offenbach
  - RED-Institut GmbH, Oldenburg
  - Universitätsklinikum Regensburg, Regensburg
  - Klinische forschung Schwerin GmbH, Schwerin
  - Studienzentrum Herzklinik Ulm MVZ, Ulm
  - Evangelisches Krankenhaus Witten, Witten
- Greece (11):
  - Evangelismos General Hospital of Athens, Athens
  - Athens Medical Center - Psychikon branch, Athens
  - University General Hospital of Heraklion, Heraklion
  - University Hospital of Ioannina, Ioannina
  - General Hospital of Nikaia-Piraeus "Agios Panteleimon", Nikaia Piraeus
  - University Hospital of Patras, Pátrai
  - G. Gennimatas General Hospital of Thessaloniki, Thessaloniki
  - AHEPA University General Hospital of Thessaloniki, Thessaloniki
  - Euromedica General Clinic of Thessaloniki, Thessaloniki
  - Ippokrateio General Hospital of Thessaloniki, Thessaloniki
  - European Interbalkan Medical Center, Thessaloniki
- Hungary (11):
  - Óbudai Egészségügyi Centrum, Budapest
  - Semmelweis Egyetem, Budapest
  - Gottsegen György Országos Kardiovaszkuláris Intézet, Budapest
  - Semmelweis University, Budapest
  - Cardiogeneral Egészségügyi Kft., Budapest
  - Medifarma 98 Kft, Nyíregyháza
  - Arina Trial Research, Orosháza
  - CoroMed, Pécs
  - KomplexLabor Diagnosztika, Szeged
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ, Szeged
  - Vita Verum Medical Egeszsegugyi Szolgaltato, Székesfehérvár
- India (13):
  - KLES Dr. Prabhakar Kore Hospital & M.R.C, Belagavi
  - Belagavi Institute of Medical Sciences - Belagavi, Belgavi
  - Eternal Heart Care Center and Research Institute, Jaipur
  - K care Hospital, Kanpur
  - Government Medical College - Kozhikode, Kozhikode
  - King George's Medical University, Lucknow
  - Sanjay Gandhi Post Graduate Institute of Medical Sciences, Lucknow
  - Kingsway Hospitals (Best Multispeciality Hospital in Nagpur), Nagpur
  - Vijan Hospital & Research Centre, Nashik
  - G.B. Pant Institute of Postgraduate Medical Education & Research, New Delhi
  - Sir Ganga Ram Hospital, New Delhi
  - All India Institute of Medical Sciences, Raipur
  - Ashirwad Hospital and Research Centre, Ulhasnagar
- Italy (16):
  - Ospedale Cazzavillan di Arzignano, Arzignano
  - Ospedale di Baggiovara, Baggiovara
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola, Bologna
  - Azienda Ospedaliera di Caserta Sant' Anna e San Sebastiano, Caserta
  - Azienda Ospedaliero Universitaria S.Anna, Ferrara
  - Azienda Ospedaliero Universitaria S.Anna, Ferrara (Cona)
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Ospedale San Martino, Genova
  - Centro Cardiologico Monzino, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Ospedale San Raffaele, Milan
  - Azienda Ospedale - Università Padova, Padua
  - A.O.U. Policlinico Paolo Giaccone, Palermo
  - Hospital Santa Maria della Misericordia in Perugia, Perugia
  - Fondazione G. Monasterio, Pisa
  - Azienda Ospedaliera Sant'Andrea, Rome
- Japan (64):
  - Akita University Hospital, Akita
  - Yamasaki Family Clinic, Amagasaki
  - Institute of Science Tokyo Hospital, Bunkyō
  - The Institute of Medical Science, Asahi Life Foundation, Chūōku
  - Shonan Fujisawa Tokushukai Hospital, Fujisawa
  - Tenjin Sogo Clinic, Fukuoka
  - Hamanomachi Hospital, Fukuoka
  - Fukuoka University Hospital, Fukuoka
  - Kyushu Central Hospital, Fukuoka
  - Gifu University Hospital, Gifu
  - Hachioji Diabetes Clinic, Hachioji-shi
  - Hakodate Municipal Hospital, Hakodate
  - Hiroshima Red Cross Hospital & Atomic-bomb Survivors Hospital, Hiroshima
  - Hiroshima Prefectural Hospital, Hiroshima
  - National Kohnodai Medical Center, Ichikawa
  - Nippon Medical School Chiba Hokusoh Hospital, Inzai
  - Nihon University Itabashi Hospital, Itabashiku
  - Shimane University Hospital, Izumo
  - Tenyoukai Central Clinic, Kagoshima
  - Shonan Kamakura General Hospital, Kamakura
  - Kanazawa University Hospital, Kanazawa
  - Mizonokuchi Okamoto Clinic, Kawasaki
  - Teikyo University Mizonokuchi Hospital, Kawasaki
  - Kobe University Hospital, Kobe
  - Yoshimura Clinic, Kumamoto
  - Omi Medical Center, Kusatsu
  - Toho University Ohashi Medical Center, Meguro-ku
  - Yokoi Clinic, Minoh
  - Nakamoto Internal Medicine Clinic, Mito
  - MinamiAkatsukaClinic, Mito
  - Miyazaki Medical Association Hospital, Miyazaki
  - Iwate Prefectural Central Hospital, Morioka
  - Nagasaki Harbor Medical Center, Nagasaki
  - Japan Public Health Association, Nagoya
  - Nagoya City University Hospital, Nagoya
  - Nakakinen clinic, Naka
  - Nishiyamadou Keiwa Hospital, Naka
  - International University of Health and Welfare Narita Hospital, Narita
  - Shimamura Memorial Hospital, Nerima-ku
  - Okayama Rosai Hospital, Okayama
  - Medical Research Institute KITANO HOSPITAL, PIIF Tazuke-Kofukai, Osaka
  - Osaka Keisatsu Hospital, Osaka
  - Osaka Metropolitan University Hospital, Osaka
  - Osaka General Medical Center, Osaka
  - Minamiosaka Hospital, Osaka
  - Abe Clinic, Ōita
  - Sato Hospital - Osaki, Ōsaki
  - Toho University Omori Medical Center, Ōta-ku
  - Sapporo Medical University Hospital, Sapporo
  - Medical Corporation Koshinkai - Thyroid and Diabetes Clinic Nakanoshima, Sapporo
  - Japan Community Healthcare Organization Hokkaido Hospital, Sapporo
  - Cardiovascular Hospital Of Central Japan - Kitakanto Cardiovascular Hospital, Shibukawa
  - Clinical Research Hospital Tokyo, Shinjuku-ku
  - Tokuyama Central Hospital, Shūnan
  - National Cerebral and Cardiovascular Center, Suita
  - Kagawa Prefectural Central Hospital, Takamatsu
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki
  - Tokyo Asbo Clinic, Tokyo
  - Sekino Hospital, Toshimaku
  - Tsuchiura Kyodo General Hospital, Tsuchiura
  - Medical Corporation Yuga Tsuruma Kaneshiro Diabetes Clinic, Yamato-shi
  - SHOWA Medical University Fujigaoka Hospital, Yokohama
  - Yokohama Minami Kyosai Hospital, Yokohama
  - Yokosuka City General Medical Center, Yokosuka
- Mexico (49):
  - Centro de Atencion al Diabetico Actopan, Actopan
  - Fundación Cardiovascular de Aguascalientes A.C., Aguascalientes
  - Medical Center Metas, Chihuahua City
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares, S.C., Ciudad Madero
  - Instituto de Diabetes, Obesidad y Nutricion, Cuernavaca
  - Centro Para El Desarrollo de La Medicina Y de Asistencia Medica Especializada S.C., Culiacán
  - Instituto Jalisciense de Investigacion en Diabetes y Obesidad, Guadalajara
  - Centro de Investigación Clínica y Medicina Traslacional (CIMeT), Guadalajara
  - Diseno y Planeacion en Investigacion Medica - Guadalajara - Calle Amado Nervo, Guadalajara
  - Instituto Jalisciense de Metabolismo, Guadalajara
  - Private Practice - Dr. Arechavaleta Granell Maria del Rosario, Guadalajara
  - Unidad de Investigación Clínica y Atención Médica HEPA S.C., Guadalajara
  - Virgen Cardiovascular Research SC, Guadalajara
  - Salud Cardiovascular, Guadalajara
  - Hermosillo Heart Team - Sinacor Hermosillo, Hermosillo
  - Instituto Cardiovascular de León S.C., León
  - Accelerium Clinical Research, Mazatlán
  - Centro Médico Lic. Arturo Montiel Rojas ISSEMYM, Metepec
  - Centro de Investigacion en Artritis y Osteoporosis SC, Mexicali
  - RM Pharma Specialists - Unidad Especializada en Datos, Mexico City
  - Grupo Medico Camino Sc, Mexico City
  - Centro de Investigación Clinica Chapultepec, Mexico City
  - Hospital de Jésus, I.A.P., Mexico City
  - Centro Médico Nacional Siglo XXI, Mexico City
  - Private Practice - Dr. Eduardo Julián José Roberto Chuquiure Valenzuela, Mexico City
  - Instituto Nacional de Cardiologia Ignacio Chavez, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City
  - Centro de Desarrollo Biomedico, Mérida
  - Kohler & Milstein Research S.A. De C.V., Mérida
  - Medical Care and Research SA de CV, Mérida
  - Centro Especializado En Diabetes, Obesidad Y Prevencion De Enfermedades Cardiovasculares, México
  - Accelerium Clinical Research, Monterrey
  - CEINV Salud, Monterrey
  - IMED Internal Medicine Clin Trials, Monterrey
  - Cardiolink Clin Trials, Monterrey
  - UBAM Unidad Biomedica Avanzada Monterrey, Monterrey
  - Clínica García Flores SC, Monterrey
  - Centro de investigación y control metabólico, Monterrey
  - Clinica de Enfermedades Cronicas y Procedimientos Especiales, SC, Morelia
  - Centro de Atención e Investigación Cardiovascular del Potosí, San Luis Potosí City
  - Servicios Integrales Nova de Monterrey S.A. de C.V., San Nicolás de los Garza
  - Centro Medico Zambrano Hellion, San Pedro Garza García
  - Fundación Santos y de la Garza Evía I.B.P, San Pedro Garza García
  - Scientia Investigación Clínica TJ, Tijuana
  - Medimanage Research, Tlalpan
  - Arké SMO S.A de C.V, Veracruz
  - FAICIC S. de R.L. de C.V., Veracruz
  - Integradora Multidisciplinaria Del Grijalva - Sinacor Villahermosa, Villahermosa
  - Hospital Angeles Xalapa, Xalapa
- Netherlands (19):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - EB Medical Research, Almere Stad
  - Meander Medisch Centrum, Amersfoort
  - OLVG Oost, Amsterdam
  - Amsterdam UMC, locatie AMC, Amsterdam
  - Ziekenhuis Rijnstate, Arnhem
  - Wilhelmina Ziekenhuis Assen, Assen
  - PT&R / PreCare Trial & Recruitment, Born
  - Ziekenhuis Gelderse Vallei, Ede
  - Tergooiziekenhuizen, locatie Hilversum, Hilversum
  - Ziekenhuis Bethesda, Hoogeveen
  - Leids Universitair Medisch Centrum, Leiden
  - Radboudumc, Nijmegen
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen
  - Bravis Ziekenhuis, locatie Roosendaal, Roosendaal
  - Erasmus Medisch Centrum, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
  - Maxima Medisch Centrum, locatie Veldhoven, Veldhoven
  - Albert Schweitzer Ziekenhuis, locatie Zwijndrecht, Zwijndrecht
- Poland (21):
  - Pro&Diagnostic, Bielsko-Biala
  - Centrum Medyczne "Hipokrates" S.C. Elżbieta I Grzegorz Grześk, Bydgoszcz
  - NZOZ Twoje Zdrowie EL Sp. z o. o., Elblag
  - Euromedica, Grudziądz
  - Gyncentrum sp. z o.o. NZOZ Holsamed - oddział Libero, Katowice
  - NZOZ Salvia CM, Katowice
  - Centrum Medyczne Komorniki, Komorniki
  - Centrum Medyczne Linden, Krakow
  - Medyczne Centrum Diabetologiczno Endokrynologiczno Metaboliczne DIAB-ENDO-MET, Krakow
  - Poliklinika Kardiologiczna Serce, Leszno
  - Centra Medyczne Medyceusz, Lodz
  - FutureMeds - Lodz, Lodz
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Clinical Best Solutions, Lublin
  - Private Practice - Dr. Michał Tomaszewski, Lublin
  - Uniwersytecki Szpital Kliniczny Nr 4 w Lublinie, Lublin
  - IRMED, Piotrkow Trybunalski
  - Centrum Szybkiej Diagnostyki Kardiologicznej "Kardiomed" M. Żabówka E. Żabówka, Tarnów
  - Futuremeds Targowek, Warsaw
  - 4 Wojskowy Szpital Kliniczny z Polikliniką SPZOZ, Wroclaw
  - Przychodnia FutureMeds Wrocław, Wroclaw
- Puerto Rico (3):
  - Advanced Clinical Research, LLC, Bayamón
  - Investigadores del Este, Humacao
  - Research and Cardiovascular Corp., Ponce
- Romania (24):
  - Cardioplus Center SRL, Baia Mare
  - Spitalul Clinic De Urgenta Prof Dr Agrippa Ionescu, Baloteşti
  - Centrul Medical Unirea, Brasov
  - Nicodiab, Bucharest
  - Hightech Medical Services SRL-Centrul pentru Studiul Metabolismului, Bucharest
  - Centrul Medical NutriLife, Bucharest
  - Delta Health Care, Bucharest
  - The National Institute of Diabetes, Nutrition and Metabolic Diseases "Prof. Dr. N. Paulescu", Bucharest
  - Spitalul Universitar de Urgență București, Bucharest
  - Spitalul Clinic Profesor Doctor Theodor Burghele, Bucharest
  - Diabet Med, Bucharest
  - Mat Cord Biomedica S.R.L., Buzău
  - Milena Sante, Galați
  - Diamed Obesity, Galați
  - Medical Practice SRL, Oradea
  - Clinica Korall, Satu Mare
  - Policlinica Astra Sibiu, Sibiu
  - SC Dentosim Queen SRL - Centrul Medical Diamed, Târgu Mureş
  - Centrul Medical Mediab, Târgu Mureş
  - Mediab S.R.L., Târgu Mureş
  - Private Practice - Dr. Cristian Podoleanu, Târgu Mureş
  - Spital Clinic Judetean de Urgenta Tg.Mures, Tg.Mures
  - Cabinet Medical Dr.Geru, Timișoara
  - Institutul de Boli Cardiovasculare Timișoara, Timișoara
- Slovakia (13):
  - PreMedix, Bratislava
  - Ambulancia diabetológie a porúch látkovej premeny a výživy - DIABEDA, Bratislava
  - Narodny ustav srdcovych a cievnych chorob, Bratislava
  - Nemocnica s poliklinikou Dunajska Streda, a.s., Dunajská Streda
  - Nemocnica s poliklinikou Sv. Lukasa Galanta, a. s., Galanta
  - Cardio D&R, Košice
  - MediVet s.r.o., Malacky
  - Nemocnica Malacky, Malacky
  - Nemocnica s poliklinikou Stefana Kukuru Michalovce a.s., Michalovce
  - BENIMED s.r.o. Kardiologicka ambulancia, Piešťany
  - Vseobecna nemocnica Rimavska Sobota, Rimavská Sobota
  - Nemocnica s poliklinikou Spišská Nová Ves, Spišská Nová Ves
  - Vranovska Nemocnica, Vranov nad Topľou
- South Korea (12):
  - Daegu Catholic University Medical Center, Daegu
  - Chosun University Hospital, Gwangju
  - Gachon University Gil Medical Center, Namdong-gu
  - Seoul National University Bundang Hospital, Seongnam
  - Korea University Anam Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - The Catholic University Of Korea St. Vincent's Hospital, Suwon
  - Ulsan University Hospital, Ulsan
- Spain (43):
  - CHUAC-Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital San Rafael - La Coruña, A Coruña
  - Parc de Salut Mar - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - EAP Osona Sud - Alt Congost S.L.P, Centelles
  - Hospital Universitario Reina Sofia, Córdoba
  - Complejo Hospitalario Universitario de Ferrol (CHUF)- Hospital Naval, Ferrol
  - Hospital Universitario Virgen Nieves, Granada
  - Hospital Infanta Elena, Huelva
  - Hospital Universitario de Jaen, Jaén
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria
  - Complejo Asistencial Universitario de León - Hospital de León, León
  - FutureMeds - Madrid, Madrid
  - Complejo Hospitalario Ruber Juan Bravo, Madrid
  - Hospital La Princesa, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Quirón Málaga, Málaga
  - H.R.U Málaga - Hospital General, Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitari Son Espases, Palma
  - CHOP - Hospital Universitario Montecelo, Pontevedra
  - Centro de Salud San Juan de la Cruz, Pozuelo de Alarcón
  - Salut Sant Joan de Reus-Baix Camp (Edp), Reus
  - Hospital Virgen del Camino, Sanlúcar de Barrameda
  - Hospital Universitario Marqués de Valdecilla, Santander
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela
  - Hospital General de Segovia, Segovia
  - Clínica nuevas Tecnologías en Diabetes y Endocrinología (NTDE), Seville
  - Hospital Quiron Infanta Luisa, Seville
  - FutureMeds - Sevilla, Seville
  - Hospital Universitario Virgen Del Rocio, Seville
  - Vithas Hospital Sevilla, Seville
  - Hospital Universitario de Toledo, Toledo
  - Hospital Clinico de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Vithas Valencia 9 de octubre, Valencia
  - Hospital Universitario Rio Hortega, Valladolid
  - Hospital Virgen de las Montañas, Villamartín
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (11):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao Sung Dist
  - National Cheng-Kung Uni. Hosp., Tainan
  - Chi Mei Medical Center, Tainan
  - National Taiwan University Hospital, Taipei
  - Cathay General Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- United Kingdom (20):
  - South Eastern Health and Social Care Trust, Belfast
  - Layton Medical Centre, Blackpool
  - Glan Clwyd Hospital, Bodelwyddan
  - Bradford on Avon Health Centre, Bradford-on-Avon
  - Bristol Royal Infirmary, Bristol
  - Panthera Biopartners - North London, Enfield
  - FutureMeds Glasgow - CPS Research, Glasgow
  - Velocity Clinical Research, High Wycombe, High Wycombe
  - HMC Health Group - Meadows Centre for Health, Hounslow
  - Raigmore Hospital, Inverness
  - Oak Tree Surgery, Liskeard
  - FutureMeds - London, London
  - The Adam Practice, Poole
  - Panthera Biopartners - Preston, Preston
  - Panthera Biopartners - Manchester, Rochdale
  - Panthera Biopartners - Sheffield, Sheffield
  - FutureMeds Teesside - Middlefield Centre, Stockton-on-Tees
  - Rame Group Practice, Torpoint
  - Sandwell General Hospital, West Bromwich
  - Panthera Clinic - York, York

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: Assessing the Impact of Muvalaplin on Major Cardiovascular Events in Adults With Elevated Lipoprotein(a) ( MOVE-Lp(a) ) — https://trials.lilly.com/en-US/trial/649436